CLINICAL TRIAL: NCT00036660
Title: A Phase II Study of SarCNU (NSC 364432) in Patients With Malignant Glioma
Brief Title: SarCNU in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I142; CAN-NCIC-IND142 (Other: PDQ); CDR0000068652 (Other: PDQ)
Record Dates: First submitted 2002-05-13; First posted 2003-07-08 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — 2-((((2-chloroethyl)nitrosoamino)carbonyl)amino)propanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: SarCNU

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of sarCNU in treating patients who have recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of SarCNU, in terms of objective response and duration of response, in patients with recurrent malignant gliomas.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.
* Determine the time to progression and survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral SarCNU on days 1, 5, and 9. Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma

  * Anaplastic astrocytoma (AA) OR
  * Glioblastoma multiforme (GBM)
* Recurrent or progressive disease by contrast-enhanced CT scan or MRI after primary surgery and radiotherapy
* At least 1 bidimensionally measurable lesion

  * At least 1 cm by 1 cm on contrast-enhanced CT scan or MRI

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm3
* Platelet count at least 120,000/mm3

Hepatic:

* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Pulmonary:

* DLCO at least 70% of predicted
* FVC at least 70% of predicted

Other:

* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix
* No ongoing or active uncontrolled infection
* No other serious illness or medical condition that would preclude study
* No history of significant neurologic or psychiatric disorder that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 6 weeks since prior immunotherapy
* No concurrent immunotherapy

Chemotherapy:

* At least 6 weeks since prior chemotherapy
* No more than 1 prior adjuvant chemotherapy regimen for AA
* No prior chemotherapy for recurrent disease
* No other concurrent chemotherapy

Endocrine therapy:

* Patients must be on a stable dose of steroids for at least 2 weeks prior to study

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No prior radiotherapy for recurrent disease
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Prior surgery for recurrent disease (e.g., stereotactic biopsy or partial resection) allowed
* At least 4 weeks since prior surgery (except for biopsy)

Other:

* At least 6 weeks since prior investigational agents
* No other concurrent investigational agents
* No other concurrent anticancer treatment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-01-10 (Actual); Primary Completion 2003-04-15 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C. Panasci, MD, Study Chair — Jewish General Hospital
Locations (5):
- Canada (5):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Webster M, Cairncross G, Gertler S, Perry J, Wainman N, Eisenhauer E. Phase II trial of SarCNU in malignant glioma: unexpected pulmonary toxicity with a novel nitrosourea: a phase II trial of the national cancer institute of canada clinical trials group. Invest New Drugs. 2005 Dec;23(6):591-6. doi: 10.1007/s10637-005-1761-3. PMID 16034522